CLINICAL TRIAL: NCT00021476
Title: Preventing Chronic Whiplash Pain: Biobehavioral Approach
Brief Title: Preventing Chronic Whiplash Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dennis Turk, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: R01AR047298 (NIH); R01AR047298 (NIH); NIAMS-064
Record Dates: First submitted 2001-07-16; First posted 2001-07-18 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Whiplash Injuries
Keywords: Whiplash; Chronic pain; Motor vehicle accidents
MeSH Terms: conditions — Whiplash Injuries; Chronic Pain | interventions — Behavior Therapy; Physical Therapy Modalities

INTERVENTIONS:
Behavioral: Behavioral treatments
Behavioral: Physical therapy

SUMMARY:
This study is aimed at developing ways to prevent acute pain from becoming chronic pain--specifically, pain associated with whiplash-associated disorders (WADs) from motor vehicle accidents. Research on the development of chronic pain due to musculoskeletal injury suggests that a person's initial emotional reactions, particularly fear of reinjury and subsequent avoidance of activity, contribute significantly to chronic pain and persistent disability. This study will treat people with WADs during the first three months after a motor vehicle accident with a behavioral and physical exercise program designed to encourage activity and discourage continued fear of movement, pain, and disability. The study will compare the effectiveness of two anxiety-reduction treatments to standard care in reducing pain and activity limitations in people with WADs in the 2 to 3 months after motor vehicle accidents.

DETAILED DESCRIPTION:
More than 1.8 million people in the United States suffer from chronic pain and disability following motor vehicle accidents (MVAs) each year. The majority of these cases start with a relatively minor neck injury. The Quebec Task Force Study on Whiplash Associated Disorders (WAD) was created in 1989 to determine the clinical, public health, social, and financial determinants of WAD. Multiple studies have described the clinical features of WAD, which include neck, shoulder, arm, low back, and head pain; tinnitus; visual symptoms; dizziness; temporomandibular joint pain; and paraesthesias. Onset of these symptoms after the injury is usually delayed for several hours and worsens within 24 to 48 hours. Neck pain is the most frequent symptom, and between 14% and 42% of patients with WAD develop chronic neck pain symptoms. Studies suggest that the neck pain will either resolve in the first few months or persist indefinitely. One variable that may predict outcome after an MVA is the acute emotional response immediately after the MVA.

A severe emotional reaction accompanied by neck pain and stiffness after an MVA could lead an injured person to avoid subsequent physical activity through such mechanisms as fear avoidance and fear of reinjury. Research investigating the evolution of chronic pain due to musculoskeletal injury suggests that initial emotional reactivity, particularly fear of reinjury and subsequent activity avoidance, contributes significantly to unremitting pain and persistent disability. Research based on this model has shown that early interventions targeting normalization of excessive emotionality and restriction of activities associated with fear following injury effectively prevent chronic pain due to back injury. No previous study has sought to intervene during the first three months after an MVA with a behavioral and physical exercise program to encourage activity and discourage continued fear of movement, pain and disability.

This study consists of two primary components: (1) To compare the effectiveness of two anxiety-reduction treatments with standard care in reducing pain and activity limitations in patients with WADs 2 to 3 months following MVAs. (2) To test whether psychological responses to the initial trauma, such as fear avoidance, fear of injury, and negative affectivity, discriminate between symptomatic WAD patients and WAD sufferers whose symptoms had resolved 2 to 3 months post-MVA.

ELIGIBILITY:
Inclusion Criteria:

* Have whiplash injury following a motor vehicle accident in the prior 4 to 10 weeks

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Pain | Measured 3 months after the accident
Functional activity | Measured 3 months after the accident
Mood | Measured 3 months after the accident

SECONDARY OUTCOMES:
Fear avoidance | Measured 3 months after the accident
Range of motion/strength | Measured 3 months after the accident
Physical symptoms | Measured 3 months after the accident

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C. Turk, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Robinson JP, Theodore BR, Dansie EJ, Wilson HD, Turk DC. The role of fear of movement in subacute whiplash-associated disorders grades I and II. Pain. 2013 Mar;154(3):393-401. doi: 10.1016/j.pain.2012.11.011. Epub 2012 Dec 1. PMID 23318127